CLINICAL TRIAL: NCT05942911
Title: A Phase II, Blinded, Randomised, Placebo Controlled Clinical Trial to Determine the Safety and Effect on Pain and Function According to RAPID-3 of IHL-675A in Patients With Rheumatoid Arthritis
Brief Title: Safety and Effect on Pain and Function According to RAPID-3 of IHL-675A in Patients With Rheumatoid Arthritis
Acronym: CHAPPII
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study suspended due to recruitment challenges not feasible to overcome
Sponsor: Incannex Healthcare Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IHL675ARAPhII
Record Dates: First submitted 2023-05-15; First posted 2023-07-12 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; MRI; RA; Rheumatoid Arthritis; Pain; Fatigue; RAMRIS; RAPID-3; Cannabidiol; CBD; Hydroxychloroquine; HCQ; Placebo; IHL-67A; Incannex; Joint pain; Stiffness
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Pain; Fatigue; Arthralgia | interventions — Cannabidiol; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IHL-675A (Experimental): 150 mg CBD, 200 mg HCQ: two soft gel capsules each containing 75 mg CBD and 100 mg HCQ twice per day for a total daily dose of 300 mg CBD and 400 mg HCQ
  Interventions: Drug: IHL-675A
- Cannabidiol (Active Comparator): 150 mg: two capsules each containing 75 mg CBD twice per day for a total daily dose of 300 mg CBD
  Interventions: Drug: Cannabidiol
- Hydroxychloroquine (Active Comparator): 200 mg: two capsules each containing 100 mg HCQ twice per day for a total daily dose of 400 mg HCQ
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Two capsules twice per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IHL-675A — Combination product containing CBD and HCQ UniGel™ technology by ProCaps®. IHL-675A consists of a solid, film coated HCQ tablet that is contained within a CBD oil solution gel cap. Each IHL-675A gel cap contains 75 mg of CBD and 100 mg HCQ.
  Arms: IHL-675A
Drug: Cannabidiol — Formulated using UniGel™ technology by ProCaps®. The CBD soft gel capsules contain 75 mg CBD oil solution. These capsules look identical to the IHL-675A UniGel™ capsules, to aid double-blinding
  Other Names: CBD; Epidiolex; Epydiolex
  Arms: Cannabidiol
Drug: Hydroxychloroquine — Formulated using UniGel™ technology by ProCaps®. The soft gel capsules each contain a 100 mg HCQ tablet. These capsules look identical to the IHL-675A UniGel™ capsules to aid double-blinding.
  Other Names: HCQ; Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo — Formulated using UniGel™ technology by ProCaps®. The soft gel capsules contain the inactive ingredients of the IHL-675A capsules and no active ingredients. These capsules look identical to the IHL-675A UniGel™ capsules to aid double-blinding.
  Arms: Placebo

SUMMARY:
The goal of this randomised, double-blind, placebo-controlled Phase II clinical trial is to assess the safety and effect of of IHL-675A in rheumatoid arthritis patients on pain, and function according to RAPID-3.

128 volunteers will be enrolled and randomised to one of four treatments (32 subjects per treatment). Each treatment will be self-administered twice daily for 24 weeks.

The four treatments are:

* Treatment 1 - IHL-675A
* Treatment 2 - CBD
* Treatment 3 - HCQ
* Treatment 4 - Placebo

DETAILED DESCRIPTION:
This is a Phase II, double-blind, randomised, placebo-controlled clinical trial to assess the safety and effect of IHL-675A (a combination of cannabidiol (CBD) and hydroxychloroquine (HCQ)) on pain and function using the RAPID-3 patient reported outcome (PRO) in patients with Rheumatoid Arthritis. This study will compare IHL-675A to the component drugs, CBD and HCQ, as well as a placebo. The study will aim to enrol a total of 128 subjects across the 4 treatment groups (32 per group).

The study will also assess structural changes in joint damage in an MRI sub-study using the Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS).

During the 28-day screening period, subjects will provide information on their demographics, medical history, history of inflammatory conditions and weight/body mass index (BMI). A physical exam, vital signs, and 12-lead ECG will be conducted. Urine and blood samples will be collected for urinalysis, to assess for pregnancy, the presence of illicit drugs and to detect any clinically significant outcomes that would exclude subjects from being eligible for the clinical trial and to measure erythrocyte sedimentation rate (ESR) and C-reactive protein (CRP) levels. A series of questionnaires will be conducted to assess eligibility and mental health status.

These questionnaires will be:

* RAPID-3
* JC 66/68
* Health Assessment Questionnaire-Disability Index (HAQ-DI)
* Columbia-Suicide Severity Rating Scale (C-SSRS) Subjects will also undergo an optical coherence tomography (OCT) eye examination to rule out retinopathy.

Subjects who have consented to the MRI sub-study will also undergo an MRI during screening.

Once the participant is deemed eligible to be enrolled in the study, the baseline visit will be performed and the participant will be randomised into one of the four treatment groups:

* Treatment 1 - IHL-675A (150 mg CBD, 200 mg HCQ: two soft gel capsules each containing 75 mg CBD and 100 mg HCQ twice per day for a total daily dose of 300 mg CBD and 400 mg HCQ)
* Treatment 2 - CBD (150 mg: two capsules each containing 75 mg CBD twice per day for a total daily dose of 300 mg CBD)
* Treatment 3 - HCQ (200 mg: two capsules each containing 100 mg HCQ twice per day for a total daily dose of 400 mg HCQ)
* Treatment 4 - Placebo (two capsules twice per day).

Subjects will visit the clinic on Day 1 and undergo baseline assessments, including:

* RAPID-3
* JC 66/68
* ACR20
* CDAI-RA
* FACIT-F
* HAQ-DI
* AE
* Concomitant medication review
* Weight/BMI
* Physical exam
* Vitals
* ECG
* Safety blood collection

Subjects will then be supplied with their first 28-day supply of their allocated treatment and will be set up with and instructed on the use of an electronic patient reported outcome (ePRO) either web based or using an app on the subject's personal device. The ePRO will be used daily by the subject to record pain, joint stiffness, tiredness, and use of other pain medication for the control of pain associated with arthritis.

Every 4 weeks, subjects will return to the clinical to undergo the same assessments and to receive the next 28-day supply of their allocated treatment. At 24 weeks, subjects will take their final dose prior to their return to the clinical for the final time (and will not receive another supply of the treatment) where they will undergo the same assessments as well as a final OCT eye exam, and subjects in the MRI sub-study will undergo a final MRI.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in the study if they satisfy all the following criteria:

1. Must have given written informed consent, before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects
2. Has been diagnosed with RA and on stable treatment for RA for at least 3 months prior to the screening visit
3. Subject has a RAPID-3 score of >4.5 at screening
4. Male or female, aged 18 or older inclusive at the screening visit
5. Body mass index (BMI) of 18 to 32 kg/m2, inclusive, at screening
6. Has at least two swollen or tender joints on the JC 66/68 at screening
7. Subject is otherwise medically healthy (in the opinion of the investigator), as determined by pre-study medical history and without clinically significant abnormalities including:

   1. Physical examination at screening without any additional clinically relevant findings apart from those consistent with RA in the opinion of the investigator.
   2. Systolic blood pressure at screening in the range of 90 to 160 mmHg and diastolic blood pressure in the range of 50 to 95 mmHg after 5 minutes in supine or semi-supine position.
   3. Pulse rate at screening in the range of 45 to 100 beats/minute after 5 minutes rest in supine or semi-supine position.
   4. Body temperature (tympanic) at screening between 35.5°C and 37.5°C.
   5. Electrocardiogram (ECG) at screening without clinically significant abnormal findings including QT interval corrected for Fredericia (QTcF) ≤470msec for females and ≤450msec for males.
8. Physically well, in the opinion of the investigator, with no severe psychiatric, cardiac, renal, endocrine, gastrointestinal, bleeding, thyroid, cholesterol, or hypertension disorders
9. Male subjects must:

   1. Agree not to donate sperm from the time of signing consent until at least 340 days (t1/2 *5 +90 days) after the last dose of study drug
   2. If engaging in sexual intercourse with a female partner who could become pregnant, must agree to use adequate contraception (defined as use of a condom plus a highly effective method of contraception (Appendix 10) from the time of signing consent until at least 340 days after the last dose of study drug).
   3. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, must agree to use a condom from the time of signing consent until at least 340 days after the last dose of study drug.
10. Female subjects must be of non-childbearing potential i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone (FSH) level consistent with postmenopausal status, per local laboratory guidelines), or, if of childbearing potential (Women who have been surgically sterilised through tubal ligation are permitted to participate, if they agree to use an additional barrier method of contraception from one month prior to the first dose of study drug, until at least 280 days (t1/2 * 5 +30 days) after the last dose of study drug.):

    1. Must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to administration of the first dose of study drug. Note: subjects must also have a negative urine pregnancy test at each clinic visit.
    2. Must agree not to donate ova or attempt to become pregnant from the time of signing consent until at least 280 days after the last dose of study drug.
    3. If not exclusively in a same-sex relationship, must agree to use adequate contraception (which is defined as use of a condom by the male partner combined with use of a highly effective method of contraception (Appendix 10) from one month prior the first dose of study drug until at least 280 days after the last dose of study drug).
11. Able to avoid strenuous exercise from 72 hours prior to each visit to the clinical unit
12. Fluent in written and spoken English
13. Willing and able to comply with all study required tasks, including the completion of questionnaires, and to adhere to the study schedule and restrictions, as instructed by the protocol.

Exclusion Criteria:

Subjects will be excluded from the study if there is evidence of any of the following at screening.

Subjects will be excluded from the study if there is evidence of any of the following at screening.

1. Known hypersensitivity to any of the study drug ingredients (cannabis products, sesame oil, hydroxychloroquine or chloroquine)
2. History of any clinically significant (in the opinion of the investigator) disorder within the last 3 months including cardiovascular (cardiac disease or arrythmias), haematologic, pulmonary, hepatic, renal, or gastrointestinal (such as cholecystitis, Gilbert's syndrome) disorders, or connective tissue, uncontrolled endocrine/metabolic, oncologic (within the last 5 years), neurologic, or any disorder within the last 3 months that may prevent the successful completion of the study or influence the absorption, distribution, metabolism, excretion or action of the study drug (in the opinion of the investigator). Note: a history of fully resolved childhood asthma is not exclusionary; a history of cholecystectomy is not exclusionary
3. Family history of QT issues
4. Currently taking or have taken hydroxychloroquine, chloroquine or any drugs containing HCQ or chloroquine within 3 months of screening
5. Taking more than 10 mg prednisone per day
6. Pregnant, lactating, planning to become pregnant
7. Known substance abuse or medical, psychological, or social conditions or significant psychiatric illness (defined as hospitalisation), suicidal ideation, or suicidal attempts that, in the opinion of the investigator, may interfere with the subjects inclusion in the clinical study or evaluation of the clinical study results
8. Regular consumption of >10 standard alcoholic drinks/week where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc/Vol], 100 mL wine [12% Alc/Vol], 30 mL spirit [40% Alc/Vol])
9. Positive urine illicit drug test at screening
10. C-SSRS score ≥4 OR reported suicidal behaviour within the past 3 months
11. Hepatic or renal impairment or disease defined as aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) >1.5 x upper limit of normal (ULN), estimated glomerular filtration rate (eGFR) <60 at screening
12. Subject has retinopathy or history thereof (as determined by the OCT eye examination at screening)
13. A positive test result for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the screening visit.
14. History of gastrointestinal disorders which may impact absorption, distribution, metabolism and/or excretion of the IP (such as cholecystitis, cholecystectomy, Gilbert's syndrome)
15. Participation in another clinical trial of an investigational drug within 30 Days or 5 half-lives of the investigational drug (whichever is longer) prior to screening
16. Any other condition or prior therapy that in the opinion of the Investigator (or delegate) would make the subject unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

MRI Sub-Study Inclusion Criteria:

Subjects may also participate in the MRI Sub-Study based on the below inclusion criteria.

1. Must have given written informed consent to participate in the MRI sub-study
2. Able and willing to undergo an MRI
3. Have at least 1 swollen and/or tender joint in left or right wrist or hand
4. Have a RAMRIS synovitis score of at least 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Change in pain and function | 24 weeks
  Routine Assessment of Patient Index Data 3 (RAPID-3) questionnaire to assess pain and function in arthritis patients.
  RAPID-3 is a pooled index of the 3 patient-reported American College of Rheumatology RA Core Data Set measures: function, pain, and patient global estimate of status. Each of the 3 individual measures is scored 0 to 10, for a total of 30. Disease severity may be classified on the basis of RAPID3 scores: >12 = high; 6.1-12 = moderate; 3.1-6 = low; < or =3 = remission

SECONDARY OUTCOMES:
Safety and tolerability - Incidence of the use of concomitant medications for pain management | 4, 8, 12, 16, 20 and 24 weeks
  Incidence of the use of concomitant pain medications for the treatment of arthritis related pain. Subjects will report the use of rescue pain medication for pain associated with arthritis using an electronic patient reported outcome (ePRO) on their personal device.
Safety and tolerability - Vital signs - Temperature | 4, 8, 12, 16, 20 and 24 weeks
  Change from baseline in body temperature (°C)
Safety and tolerability - Vital signs - Pulse Rate | 4, 8, 12, 16, 20 and 24 weeks
  Change from baseline in pulse rate (BPM)
Safety and tolerability - Vital signs - Respiratory Rate | 4, 8, 12, 16, 20 and 24 weeks
  Change from baseline in respiratory rate (RPM)
Safety and tolerability - Vital signs - Blood Pressure | 4, 8, 12, 16, 20 and 24 weeks
  Change from baseline in systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) to report change in blood pressure
Safety and tolerability - 12-lead ECG | 4, 8, 12, 16, 20 and 24 weeks
  Change from baseline in 12-lead ECG results: PR interval, QRS, QTcF
Safety and tolerability - Adverse Events | 4, 8, 12, 16, 20 and 24 weeks
  Assess the number of treatment emergent adverse events (TEAEs) and serious treatment emergent adverse events associated with the dosing of IHL-675A in comparison to the active comparators (CBD and HCQ), and placebo.
Safety and tolerability - OCT Eye Exam | 24 weeks
  Changes from baseline in retinopathy as assessed by Optical Coherence Tomography (OCT) eye exam
Safety and tolerability - The Columbia Suicide Severity Rating Scale (C-SSRS) | 24 weeks
  Change from baseline in suicidality assessed by The Columbia Suicide Severity Rating Scale (C-SSRS). The C-SSRS is an instrument that measures suicidal ideation and behaviour. The ideation subscale evaluates severity on a 5-point scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The behaviour subscale assesses various categories of suicidal behaviour. Higher scores on the C-SSRS represent more severe levels of suicidal ideation or behaviour. Lower scores, therefore, indicate a better outcome as it represents lower levels of suicidal ideation or behaviour.
Change in pain - Routine Assessment of Patient Index Data 3 (RAPID-3) | 4, 8, 12, 16 and 20 weeks
  Change in pain from baseline. Assessed by change in Routine Assessment of Patient Index Data 3 (RAPID-3) score relative to baseline. RAPID-3 is a composite score that measures physical function, pain, and patient global assessment on a scale from 0 to 30, with higher scores indicating worse outcomes (i.e., more pain and disability). A decrease in the RAPID-3 score from baseline represents an improvement.
Change in fatigue - Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | 4, 8, 12, 16, 20 and 24 weeks
  Change in fatigue from baseline. Assessed by change in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score. FACIT-F is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function on a scale from 0 to 160. Higher scores indicate better outcomes (i.e., less fatigue). An increase in the FACIT-F score from baseline represents an improvement.
Change in quality of life - Health Assessment Questionnaire - Disability Index (HAQ-DI) | 4, 8, 12, 16, 20 and 24 weeks
  Change in quality of life from baseline. Assessed by change in Health Assessment Questionnaire - Disability Index (HAQ-DI) score. The HAQ-DI assesses a patient's level of functional ability on a scale from 0 to 3. Higher scores indicate worse outcomes (i.e., greater disability). A decrease in the HAQ-DI score from baseline represents an improvement.
Change in disease activity - ACR20 | 4, 8, 12, 16, 20 and 24 weeks
  Change in disease activity from baseline. Assessed by change in American College of Rheumatology-20 (ACR20) response rate. The ACR response is scored as a percentage improvement, comparing disease activity at two discrete time points (usually baseline and post-baseline comparison). ACR20 is ≥ 20% improvement
Change in disease activity - JC66/68 | 4, 8, 12, 16, 20 and 24 weeks
  Change in disease activity from baseline. Assessed by change in joint swelling/tenderness count 66/68 (JC66/68). The 66/68 Joint Count evaluates 66 joints for swelling and 68 joints for tenderness and pain with movement. Note that the hip joints can be evaluated for tenderness only-not for swelling. The total score is composed of points that are based on the presence of pain and/or swelling in a joint
Change in disease activity - CDAI-RA | 4, 8, 12, 16, 20 and 24 weeks
  Change in disease activity from baseline. Assessed by change in clinical disease activity index for rheumatoid arthritis (CDAI-RA) score. CDAI is based on the simple summation of the count of swollen/tender joint count of 28 joints along with patient and physician global assessment on VAS (0-10 cm) Scale for estimating disease activity. The CDAI has range from 0 to 76.
Change in inflammatory serology - C-Reactive Protein (CRP) | 4, 8, 12, 16, 20 and 24 weeks
  Change in CRP levels from baseline. Assessed by the change in blood C-reactive protein (CRP) levels relative to baseline. CRP is a systemic marker of inflammation. The measurement is reported in milligrams per litre (mg/L). Higher levels of CRP typically indicate a higher level of systemic inflammation, so a decrease in CRP levels from baseline would generally indicate an improvement.
Change in inflammatory serology - Erythrocyte sedimentation rate (ESR) | 4, 8, 12, 16, 20 and 24 weeks
  Change in ESR levels from baseline. This outcome is assessed by the change in blood erythrocyte sedimentation rate (ESR) levels relative to baseline. ESR is a systemic marker of inflammation. The measurement is reported in millimetres per hour (mm/hr). Higher ESR levels typically indicate a higher level of systemic inflammation, so a decrease in ESR levels from baseline would generally indicate an improvement.
Change in tiredness | 24 weeks
  Change in tiredness from baseline. Assessed by an electronic patient reported outcome (ePRO). Subjects will be prompted daily to answer a set of 5 questions that will ask the patient about their pain, joint stiffness duration and severity, and tiredness, and to record the use of any concomitant medication for pain associated with arthritis.
Change in pain (daily) | 24 weeks
  Change in pain from baseline. Assessed by an electronic patient reported outcome (ePRO). Subjects will be prompted daily to answer a set of 5 questions that will ask the patient about their pain, joint stiffness duration and severity, and tiredness, and to record the use of any concomitant medication for pain associated with arthritis.
Change in joint stiffness duration | 24 weeks
  Change in joint stiffness duration from baseline. Assessed by an electronic patient reported outcome (ePRO). Subjects will be prompted daily to answer a set of 5 questions that will ask the patient about their pain, joint stiffness duration and severity, and tiredness, and to record the use of any concomitant medication for pain associated with arthritis.
Change in joint stiffness severity | 24 weeks
  Change in joint stiffness severity from baseline. Assessed by an electronic patient reported outcome (ePRO). Subjects will be prompted daily to answer a set of 5 questions that will ask the patient about their pain, joint stiffness duration and severity, and tiredness, and to record the use of any concomitant medication for pain associated with arthritis.
Effect of IHL-675A on cytokines | 12 and 24 weeks
  Change in cytokines IL-1β, IL-6, TNF levels compared to pre-dose levels.

OTHER OUTCOMES:
Structural effects of IHL-675A | 24 weeks
  Change in Rheumatoid Arthritis Magnetic Resonance Imaging Score (RAMRIS) at 24 weeks (visit week 25) compared to baseline in a sub-study of subjects who have affected wrist and metacarpophalangeal joints (applicable to sub-study only).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hall, Prof., Principal Investigator — Emeritus Research
Locations (10):
- Australia (10):
  - Paratus Clinical (Woden Dermatology), Phillip, Australian Capital Territory
  - Genesis Research Services, Broadmeadow, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Novatrials, Kotara, New South Wales
  - Emeritus Research, Sydney, New South Wales
  - Coast Joint Care, Maroochydore, Queensland
  - AusTrials Westside (Taringa), Taringa, Queensland
  - AusTrials Wellers Hill, Wellers Hill, Queensland
  - Emeritus Research Melbourne, Camberwell, Victoria
  - Captain Sterling Medical Centre, Nedlands, Western Australia